CLINICAL TRIAL: NCT07247461
Title: TOLA: Transthoracic Drainage of Lung Abscesses. A National Randomized Trial
Brief Title: Transthoracic Drainage of Lung Abscesses. A National Randomized Trial.
Acronym: TOLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOLA
Record Dates: First submitted 2025-10-01; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Lung Abscess
Keywords: Lung Abscess; Transthoracic drainage; Length of hospital stay; Randomized trial
MeSH Terms: conditions — Lung Abscess

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transthoracic drainage (Active Comparator): Patients in this arm will receive a Transthoracic drainage in their lung abscess in combination with standard treatment with IV antibiotics
  Interventions: Procedure: Transthoracic drainage
- Control group (No Intervention): Patients in this arm will receive standard treatment will IV antibiotics

INTERVENTIONS:
Procedure: Transthoracic drainage — Patients randomized to the intervention arm will receive a Transthoracic drain in their lung abscess.
  Arms: Transthoracic drainage

SUMMARY:
This study aims to investigate if early drainage of lung abscesses, in addition to standard antibiotic treatment, leads to shorter length of hospital stay.

Study Design

This is a randomized, controlled clinical trial. That means participants will be randomly assigned to one of two groups:

1. Drainage group: Receives a chest tube (drain) inserted through the chest wall into the abscess in combination with standard intravenous antibiotics.
2. Control group: Receives standard intravenous antibiotics only

Each participant has a 50/50 chance of being placed in either group.

During Hospital Stay All participants will begin treatment with intravenous antibiotics (piperacillin/tazobactam). If assigned to the drainage group, a trained medical team will insert a small tube into the abscess to drain the pus. The tube is flushed three times a day with sterile saline.

Participants will also:

* Fill out two short health questionnaires at the start and during follow-up.
* Have relevant medical history collected from their hospital records.
* Undergo routine scans (CT), blood tests, and lung assessments as part of standard care.
* A cheek swab will be taken from all participants to study mouth bacteria..

For those receiving drainage the pus from the lung abscess will be collected for microbiological analysis.

Microbiology samples will be stored in a research biobank and destroyed after analysis.

Follow-up after discharge

* 1 week: A phone call to check symptoms and infection levels via a blood test.
* 4 and 12 weeks later: In-person checkups at the lung clinic, including:

  * 6-minute walk test
  * Lung function test
  * Repeat health questionnaires
  * CT scan
  * Blood tests (up to 20 ml in total over the study)
* 1 years: Medical records are reviewed to asses morbidity and mortality.

Participants The study will include 84 adult patients who are hospitalized with a lung abscess larger than 4 cm, located near the outer part of the lung. Inclusion will take place at five university hospitals in Denmark

Why This Study Matters There are no official guidelines for treating lung abscesses, and research is limited. This study could offer vital new insights that help update treatment recommendations in Denmark and internationally.

Because all five Danish regions are involved, the results could quickly be implemented into daily practice, improving care for future patients with this serious condition.

DETAILED DESCRIPTION:
Trial design, setting and time frame The study is a multicentre, national, randomized controlled, open-label trial involving respiratory departments at university hospitals across all regions of Denmark. Patient enrollment is expected to to beguin early 2026 and continue for a 2-year period, concluding in early 2028.

Eligibility criteria Patients are eligible for inclusion to the study if they are above 18 years of age and admitted to the hospital with a lung abscess (LA) equal or larger than 4 cm containing fluid and in contact with the outer 1/3 of the lung.

Patients can be screened for eligibility at any hospital in Denmark. If the patient is eligible for inclusion and accepts participation in the study, the patient will be transferred to the respiratory department at the regional university hospital where randomization and inclusion will be performed.

Intervention - drainage Transthoracic drainage (TTD) will be initiated as soon as possible in the intervention group and within 72 hours of inclusion and randomization. Insertion of a drainage tube will be guided by ultrasound or computed tomography, decided by the operator case-by-case. Discontinuation of anticoagulant treatment and local anesthetics will be applied according to local guidelines. Choice of tube type (seldinger, one-step) will be decided by the operator. In cases where multiple LA are present, a tube will be placed in the largest LA accessible for drainage. If the tube is accidentally removed, indication for reinsertion will be decided by the treating physician.

The tube will be assessed daily and flushed three times daily with saline to ensure patency. Daily monitoring and documentation of chest tube input and output will be conducted, supplemented by a brief assessment of symptoms related to drainage.

Duration of drainage will be decided case-by-case by the treating physician. The following criteria are used to assist the treating physician in determining when to remove the drain:

* Clinical improvement of the patient (no fever and improved general condition).
* Paraclinical satisfactory response (decrease in leukocytes and C-reactive protein (CRP)).
* Imaging with improvement
* Drain with clear fluid by rinsing. Drainage should continue until above criteria are met. If treating physician detects complications or conditions that worsens the patients' health, they may choose to remove the drain.

The intervention group will also receive the same antibiotic treatment as the control group.

Comparator - antibiotics Patients will be treated with 4g/0.5g Piperacillin/tazobactam intravenously (IV) four times daily. The length of IV treatment is decided by the treating physician. In cases of diseases progression, allergy to specific antibiotic or microbiological findings, the treating physician can adjust the choice of antibiotics.

After the initial treatment with IV antibiotics, all patients will be switched to oral antibiotics with 500mg amoxicillin/125mg clavulanic acid. Oral treatment can be initiated when all the following criteria are meet:

* Clinical improvement (no fever and improved general condition)
* Paraclinical satisfactory response (decrease in leukocytes and CRP)
* Imaging with improvement
* Drain/pigtail is removed The length of the oral antibiotic phase will be decided by the treating physician, depending on clinical improvement, paraclinical response and radiological assessment. The treating physician can adjust the choice of oral antibiotics in case of specific bacteriological findings, drug allergies or potential drug-drug interactions.

Standard concomitant care is allowed for all patients according to national guidelines such as pain relief medication, thrombosis prophylactic, nutritional support and respiratory physiotherapy decided by treating physician.

Discharge

Treating physician decides when the patient is ready for discharge. The TTD must be removed, and the patient must be on oral antibiotics. The following criteria will be used to guide time of discharge inspired by the Danish guideline for pneumonia:

* Temperature < 37.8 degrees
* Heartrate < 100 bpm
* Systolic blood pressure >90 mmHg
* Respiratory rate < 24/minute
* Habitual mental state

Outcomes Primary outcome is length of hospital stay from admission to discharge measured in days.

Harms Safety will be evaluated case by case by rate of adverse events, device adverse reactions and complication in the form of pleural empyema, pneumothorax, bronchopleural fistula and hemothorax during admission and clinical follow-up.

Sample size The power calculation is based on clinical experience, national data and international studies. A study reported a mean length of stay of 18 days (SD 6.5) in patients treated with antibiotics. We anticipate a 25% reduction in length of hospital stay among patients treated with TTD. As the distribution of length of hospital stay is expected to be skewed, a logarithmic transformation is performed prior to calculation of sample size.

Assuming a power of 80%, a two-sided significance level of 0.05 and an expected dropout rate of 10%, 42 patients will be enrolled in each arm, yielding a total sample size of 84 participants.

Randomization and blinding Patients will be randomized 1:1 to either

1. Intervention: TTD in combination with standard antibiotic treatment.
2. Comparator: Standard antibiotic treatment alone. Randomisation will be carried out by REDCap (Research Electronic Data Capture) in blocks of 4 stratified for each region to insure equal distribution of patients and interventions.

Patients and treating healthcare staff will not be blinded. Statisticians who will perform the statistical analysis will be blinded to treatment allocation.

Data collection and follow-up During hospitalization patients will be monitored according to local practice. All data related to blood tests, radiological procedures, medical treatment, microbiological samples, and the management of the TTD will be systematically recorded in the study. A standardized template will be employed during medical rounds to ensure consistency in data collection both across consecutive days and between participating hospitals. Upon inclusion, an audit of each patient's medical record will provide information on comorbidities, prior lung function, previous radiological procedures, and relevant medical history. Additionally, patients will complete a questionnaire including COPD assessment test (CAT) and the EuroQol -5 dimensions, 5 level instrument (EQ-5D-5L) to evaluate health-related quality of life (supplementary).

Following hospital discharge, all patients will be monitored up in outpatient clinics at the respiratory departments of the regional university hospitals. Follow-up assessments will be conducted at 1, 4, and 12 weeks, focusing primarily on clinical status, biochemical parameters, and radiological resolution. One year after discharge, patients' medical records will be reviewed to evaluate morbidity and mortality.

All clinical data will be registered in a prospective REDCap database, hosted at Aarhus University with at each regional university hospital appointing a responsible investigator for data entry and oversight. The REDCap database is a secure data management system, fully compatible with all regulatory guidelines. Any physical data will be stored at the department of respiratory disease and allergy at Aarhus University Hospital

Statistical methods Results will be reported in accordance with CONSORT guidelines. Data is extracted from REDCap database and data analysis is performed using the statistical software R (4.5.2).

Data will be reported in each group as median with interquartile ranges (IQR). For the primary endpoint, length of hospital stay, defined as the number of days from admission to discharge, patients who die before discharge will be excluded from the primary analysis. A predefined sensitivity analysis will be performed to test whether death before discharge affects the primary endpoint.

Between group comparison will be performed using a t-test on log-transformed length of hospital stay to account for skewed distribution. The results will be presented as median ratios with 95% confidence intervals.

Sensitivity analysis will include time-to-discharge models (Cox proportional hazards) to assess the impact of deaths and censored observations (patient hospitalized at end-of-study or lost to follow-up). Analysis will adjust for age, gender, and pulmonary comorbidities.

Secondary outcomes will be reported as median with IQR for continuous variables and n(%) for binary outcomes. Continuous secondary outcomes will be compared using t-test or Wilcoxon rank sum test depending on distribution of data. Binary outcomes will be compared using Chi-square test for unadjusted analyses. If adjustment is required, logistic regression will be applied, and results will be reported as odds ratio with 95% confidence intervals. Repeated measurements (e.g., patient reported outcomes) will be analyzed using linear mixed model with treatment groups and time as fixed effects and patients as a random effect.

Effect of the intervention will primarily be analyzed according to intention-to-treat principles. In addition, a per protocol analysis will be conducted.

Ethics, approvals and monitoring This study is approved by the Danish Research Ethics Committee (1-10-72-146-25) and Central Region Denmark (1-16-02-539-25). Information about the subjects is protected under the EU's General Data Protections Regulation (GDPR), the Danish Personal Data Processing Act and Danish Health Act. The study will be conducted in accordance with the Helsinki II Declaration.

Since TTD is a recognized treatment for selected cases of LA the study is not categorized as test of medical equipment and monitoring by the Good Clinical Practice Unit (GCP) is not legally required. However, the study will be conducted according to GCP principles.

Patients will provide written informed consent according to Danish legislation prior to enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Signed informed consent.
* CT scan compatible with LA (one or more cavitating lesions with liquid content).
* Clinical findings suggestive of ongoing infection.
* Lung abscess size ≥ 4 cm in diameter.
* Imaging indicates that the abscess contains fluid.
* The abscess involves the outer one-third of the lung.

Exclusion Criteria:

* Pregnancy. Prior to inclusion of fertile women, a negative pregnancy test must be available.
* Brest feeding.
* Predicted survival of less than 3 months.
* Known tuberculosis or non-tuberculous mycobacteriosis.
* Known chronic pulmonary aspergillosis.
* Patients with a primary suspicion of lung cancer
* Recent (<3 months) contact with health facilities outside Scandinavia.
* Patients in whom anticoagulant treatment cannot be discontinued, or in whom the treatment pause does not allow drainage within 72 hours.
* Coagulopathy or other increased bleeding risk that cannot be corrected to allow drainage within 72 hours.
* Hemodynamic and/or respiratory unstable patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | From the patient is admitted to the hospital (day one) to the patient is discharged
  Primary outcome is length of hospital stay from admission to discharge measured in days.